CLINICAL TRIAL: NCT03722290
Title: Evaluate the Efficacy and Safety of Metformin in Children and Adults With Fragile X Syndrome: an Open-label Study
Brief Title: Metformin in Children and Adults With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: FRAXA Research Foundation (Other)
Responsible Party: Principal Investigator, Çaku, Principal Investigator, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-2797
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Fragile X Syndrome
Keywords: Metformin; Insulin signalisation
MeSH Terms: conditions — Fragile X Syndrome | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Open-label trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): Metformin 500mg twice a day per os for 9 weeks
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Oral administration of metformin 250mg (twice a day) for the 1st week followed by metformin 500mg (twice a day) for the next 8 weeks.
  Other Names: Glucophage

SUMMARY:
Fragile X Syndrome (FXS) is caused by loss of FMR1 expression on the X chromosome that leads to increased mRNA translation, which results in hyperactivation of ERK (extracellular signal-regulated kinase) and mTORC1 (mechanistic target of rifampicin complex 1) signalling and consequently in synaptic dysfunction and neurological development. There is presently no cure for FXS. Recent studies suggest that metformin (a widely prescribed drug for type II diabetes in children and adults) which crosses the blood-brain barrier, corrects various neurological and behavioral FXS phenotypes by normalizing ERK signaling, EIF4E phosphorylation and lowering expression of MMP9 to normal. Since this drug has not been previously used specifically for treatment of FXS (only few cases reported), the investigators propose an open-label trial of metformin in children and adults with FXS to better understand the safety and efficacy in both behavior and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 et 45 years old
* BMI > 18.3
* Molecular diagnosis of FXS
* Accompanied by his legal tutor

Exclusion Criteria:

* Pregnancy/Breastfeeding
* Intolerance to metformin
* History of lactic acidosis
* Gastric/renal/hepatic pathology
* Acute medical condition
* Concomitant use of ACE inhibitors
* Modification of antipsychotic treatments in the last 6 weeks

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverses events reported during the study | 9 weeks
  Number and severity of adverse events related to metformin treatment
Change from baseline in the total score of the FX-normed Aberrant Behavior Checklist-Community after 9 weeks of metformin treatment | Baseline, Week 9
  The ABC-C is a 58-item caregiver-rated behavior scale where each item ranges from 0 (not a problem) to 3 (severe problem).

SECONDARY OUTCOMES:
Level of cortical excitability using Transcranial Magnetic Stimulation (TMS) | Baseline, Week 9
  The effects of metformin on cortical excitability will be measured using a magnetic stimulation on the primary motor cortex to assess intracortical facilitation and inhibition
Level of synaptic plasticity using Electroencephalography (EEG) | Baseline, Week 9
  The effects of metformin on synaptic plasticity will be measured using the changes in amplitude of EEG waves
Changes from baseline in the score of each subscale of the Aberrant Behavior Checklist-Community (ABC-C) | Baseline, Week 9
  Determining if metformin lowers the score of each subscale of the ABC-C: Irritability (18 items), hyperactivity (10 items), lethargy (16 items), social avoidance (4 items), stereotypy (6 items) and inappropriate speech (4 items). Each item is scored from 0 (not a problem) to 3 (severe problem).
Changes from baseline in the Global Executive Composite (GEC) baseline score of the Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, Week 9
  The BRIEF is a 86-item questionary evaluating executive functions rated on a 3-point Likert scale: 1 (never), 2 (sometimes) and 3 (often).
Changes from baseline in the score of 4 subtests of the computerized cognitive Test of Attentional Performance for Children | Baseline, Week 9
  KiTAP is a computerized continuous test of attention assessing the ability to maintain attention in the presence of distractors. The 4 subtests used are Alertness reaction time, Distractibility commission errors, Go/No-Go commission errors and Flexibility errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No